CLINICAL TRIAL: NCT02476643
Title: Integrative Therapy in Gastroenterology - a Prospective Observational Trial in a Department of Internal and Integrative Medicine
Brief Title: Integrative Gastroenterology - an Observational Trial
Acronym: InteGast
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Romy Lauche, Principal Investigator, Universität Duisburg-Essen
Other Study IDs: 15-6183-BO InteGast
Record Dates: First submitted 2015-06-12; First posted 2015-06-19 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Crohns Disease; Ulcerative Colitis; Irritable Bowel Syndrome
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Integrative Therapy: This group receives and integrative therapy at the Department of Internal and Integrative Medicine, i.e. a combination of conventional diagnostic and therapeutic interventions with specific naturopathic, and complementary medicine approaches, and physical therapy.
  Patients are admitted to the hospital ward for 14 days.
  Interventions: Other: Integrative Therapy

INTERVENTIONS:
Other: Integrative Therapy — This group receives an integrative therapy at the Department of Internal and Integrative Medicine, i.e. a combination of conventional diagnostic and therapeutic interventions with specific naturopathic, and complementary medicine approaches, and physical therapy.

SUMMARY:
This study aims to test, if a two-week integrative therapy in an internal medicine ward will improve symptoms, disability and quality of life in patients with inflammatory bowel disease or irritable bowel syndrome.a It shall further be tested, if those changes are associated with attitudes and experiences towards complementary and alternative medicine, anxiety, depression and stress perception as well as body awareness and responsiveness.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* diagnosed with Irritable Bowel Syndrome (IBS) or Inflammatory Bowel Disease (IBD)
* written informed consent

Exclusion Criteria:

* participation in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients with Inflammentory Bowel Disease admitted to the Department of Internal and Integrative Medicine.
  100 patients with Irritable Bowel Syndrome admitted to the Department of Internal and Integrative Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Symptoms Severity IBS-SSS | 2 weeks
  Symptoms Severity assessed by Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) (Francis, 1997)
Symptoms Severity CAI | 2 weeks
  Symptoms Severity assessed by Clinical Activity Index (CAI) (Rachmilewitz 1989)
Symptoms Severity CDAI | 2 weeks
  Symptoms Severity assessed by Crohn Disease Activity Index (CDAI)

SECONDARY OUTCOMES:
Symptoms Severity IBS-SSS | 24 weeks
  Symptoms Severity assessed by Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) (Francis, 1997)
Symptoms Severity CAI | 24 weeks
  Symptoms Severity assessed by Clinical Activity Index (CAI) (Rachmilewitz 1989)
Symptoms Severity CDAI | 24 weeks
  Symptoms Severity assessed by Crohn Disease Activity Index (CDAI)
Disability MYMOP | 2 weeks
  Disability assessed by Measure Yourself Medical Outcome Profile (MYMOP) (Paterson 1996)
Disability MYMOP | 24 weeks
  Disability assessed by Measure Yourself Medical Outcome Profile (MYMOP) (Paterson 1996)
Quality of Life IBS-QOL | 2 weeks
  Irritable Bowel Syndrome Quality of Life measurement (IBS-QOL) (Patrick, 1998)
Quality of Life IBS-QOL | 24 weeks
  Irritable Bowel Syndrome Quality of Life measurement (IBS-QOL) (Patrick, 1998)
Quality of Life IBDQ | 2 weeks
  Inflammatory Bowel Disease Questionnaire (IBDQ) (Cooney et al., 2007)
Quality of Life IBDQ | 24 weeks
  Inflammatory Bowel Disease Questionnaire (IBDQ) (Cooney et al., 2007)
Self efficacy questionnaire SWE | 2 weeks
  Self efficacy questionnaire (SWE) (Schwarzer and Jerusalem, 1995)
Self efficacy questionnaire SWE | 24 weeks
  Self efficacy questionnaire (SWE) (Schwarzer and Jerusalem, 1995)
Body awareness BAQ | 24 weeks
  Body awareness assessed by Body Awareness Questionnaire (BAQ) (Shields et al., 1989)
Body awareness BRS | 24 weeks
  Body awareness assessed by Body Responsiveness Scale (BRS) (Daubenmier, 2005)
Adverse effects | 2 weeks
  Number of participants with any adverse effect during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof, MD, Principal Investigator — Department of Internal and Integrative Medicine, Kliniken Essen-Mitte
Locations (1):
- Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Essen, Germany